CLINICAL TRIAL: NCT05709223
Title: Feasibility, Prospective, Within-subject, Interventional Study Comparing the Performance of a Categorical Loudness Scaling Based Fitting With a Behavioural Fitting in Adults With a Nucleus Cochlear Implant in the First 3 Months Post-activation
Brief Title: Comparing the Performance of a Categorical Loudness Scaling Based Fitting With a Behavioural Fitting in Adults With a Nucleus Cochlear Implant 3 Months Post-activation
Acronym: CALOS4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Collaborators: QbD Clinical (Industry); Avania (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AI5824
Record Dates: First submitted 2022-12-01; First posted 2023-02-02 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2024-06

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Masking Description: Participants are blinded to the order of fitting method. Some participants will use first the Behavioural program followed by the investigational program while the other group will use each of these conditions in the opposite order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants receiving both Categorical Loudness Scaling Based Fitting and behavioural fitting. (Experimental): Participants will receive a categorical loudness scaling based fitting (Interventional) and behavioural fitting with 4 weeks experience of both MAPS
  Interventions: Device: Categorical loudness scaling based fitting using the Nexus Research System.; Device: Behavioural fitting using Custom Sound Suite (CSS 6.3) Software

INTERVENTIONS:
Device: Categorical loudness scaling based fitting using the Nexus Research System. — The Nexus Research system is used in combination with other devices as part of a hearing implant system. It is intended to create and modify hearing profiles, to monitor the performance of the system and to facilitate Firmware updates of the system. It is also intended to be used with other devices of a hearing implant system to make volume adjustments to the processing unit, to download pre-defined MAPs and to collect data from tests and questionnaires using a compatible device.
  Other Names: The Nexus Research System.
Device: Behavioural fitting using Custom Sound Suite (CSS 6.3) Software — The comparator is the commercially available fitting method (i.e., the behavioural measurement of active channels) using Custom Sound Suite (CSS 6.3) software

SUMMARY:
This study aims to collect data in newly implanted cochlear implant-recipients to inform future development of fitting methods to optimally and efficiently program a cochlear implant.

DETAILED DESCRIPTION:
Firstly, it aims to collect data to investigate if the new fitting method gives a good fit of MAP for newly implanted CI-recipients in terms of performance outcomes, compared to the standard streamlined behavioural fitting after 3 months of use. Secondly, it aims to collect data to further refine the new fitting method beyond what is evaluated within this study.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older (no upper age limit).
2. Post-lingually deafened defined as severe or greater sensorineural hearing loss onset after the age of 2 years as reported by the subject
3. Unilaterally implanted with the CI600 Series (CI612, CI622, CI632) or CI500 series (CI512, CI522, CI532) cochlear implant.
4. Fluent speaker in the language used to assess speech perception performance, as determined by the investigator.
5. Willingness to participate in and comply with all requirements of the protocol.
6. Willing and able to provide written informed consent

Exclusion Criteria:

1. Score below 3 on the screening subset of questions from the Mobile Device Proficiency Questionnaire.
2. Subject who will be programmed with an acoustic component in the implanted ear.
3. Pure tone average (average of unaided thresholds at 0.5, 1, 2 and 4 kHz) less than or equal to 30 dB HL and aided word score of more than 80% in the contralateral ear.
4. Diagnosis of auditory neuropathy.
5. Additional health factors, known to the investigator, that would prevent or restrict participation in the evaluations, including significant visual impairment and/or dexterity issues.
6. Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator.
7. Investigator site personnel directly affiliated with this study and/or their immediate families: immediate family is defined as a spouse, parent, child, or sibling.
8. Cochlear employees or employees of Contract Research Organizations or contractors engaged by Cochlear for the purposes of this investigation.
9. Current participation, or participation in another interventional clinical study/trial in the past 30 days, involving an investigational drug or device (unless the other investigation was/is a Cochlear sponsored investigation and determined by the investigator or Sponsor to not impact this investigation). -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
Change in Percentage of correct monosyllabic word scores in quiet (S0) at 50 dB SPL | 2 days(In booth testing)
  To determine whether the Loudness Target (LT) MAP provides non-inferior speech understanding in quiet compared to the Behavioural MAP. Percentage of correct monosyllabic word scores in quiet (S0) at 50 dB SPL averaged across the sessions at visit 4 and visit 5. Higher the score better the outcome.
Change in Adaptive sentence in noise scores (S0N0 test setup) | 2 days (In booth testing)
  To determine whether the Loudness Target (LT) MAP provides non-inferior speech understanding in noise compared to the Behavioural MAP. Adaptive sentence in noise scores (S0N0 test setup) averaged across the sessions at visit 4 and visit 5.

SECONDARY OUTCOMES:
Speech, Spatial and Qualities of Hearing Scale (SSQ12) ratings | 4 weeks
  To determine whether the LT MAP provides non-inferior speech understanding, sound quality and spatial hearing performance subjective ratings in daily life compared to the Behavioural MAP.
  The SSQ-12 is comprised of 12 items using the response format on a scale from 0 to 10, were 0 equals no ability and 10 equals perfect ability. These are divided into three sub-scales and the questions 1-5 are from the speech sub-scale, 6-8 from the spatial, and 9-12 from the qualities sub-scale. The three sub-scales are the average of the questions within. A 'not applicable' option is given for each item.
  The change between LT to Behavioural MAP is then calculated and the theoretical score could vary between -10 to + 10. The higher the score the better benefit and positive score indicates improved hearing, a negative value an impaired hearing.
Percentage correct monosyllabic word scores in quiet (S0) at 60 dB SPL | One day (in booth testing)
  To determine whether the LT MAP provides non-inferior speech understanding in quiet compared to the Behavioural MAP early post activation.
Adaptive Digit Triplet Test (DTT) in noise scores | One day (in clinic testing)
  To determine whether the LT MAP provides non-inferior speech understanding in noise compared to the Behavioural MAP early post activation. Digit triplets are presented adaptively at different SNRs to estimate a patient's Speech Reception Threshold for 50%-digit triplet identification and expressed as a dB SNR (SNR50). The SRT is determined at the end of the test. A higher SRT means a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Anke Plasmans, Study Director — Cochlear
Locations (4):
- Cochlear Americas, Lone Tree, Colorado, United States
- Australia (2):
  - Cochlear Sydney, Sydney, Sydney
  - HEARnet, Carlton, Victoria
- Medizinische Hochschule Hannover (MHH), Hanover, Hannover, Germany

IPD SHARING:
Plan to Share IPD: No